CLINICAL TRIAL: NCT03758989
Title: A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Brief Title: A Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carla Casulo, Associate Professor of Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULYM18040
Record Dates: First submitted 2018-11-15; First posted 2018-11-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: DLBCL
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Baseline PET (Experimental): R-CHOP
  Interventions: Drug: Rituximab Prednisone; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab Prednisone — A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Drug: Cyclophosphamide — A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Drug: Doxorubicin — A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Drug: Vincristine — A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma
Drug: Prednisone — A Phase II Study of PET Adapted Therapy and Non-invasive Monitoring for Previously Untreated Limited Stage Diffuse Large B Cell Lymphoma

SUMMARY:
The overarching goals of this study are to measure levels of circulating tumor DNA (ctDNA) in patients with early stage diffuse large B cell lymphoma (DLBCL), to assess the change in ctDNA during treatment in order to prospectively identify markers of treatment failure, and to use ctDNA as a future tool for response adapted therapy.

DETAILED DESCRIPTION:
The long-term objective of this proposal is to determine the correlation between FDG-PET and MRD, as measured by ctDNA in patients with early stage DLBLC.

Patients will be treated with standard chemoimmunotherapy and radiation based on the recently completed SWOG S1001 study, however no radioimmunotherapy will be used (NCT01359592). Response to treatment will be determined by contemporary Deauville criteria. Assessment of ctDNA (non-invasive disease monitoring) will be determined at diagnosis and will continue at pre-defined specific time points after therapy is complete.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated limited stage non bulky DLBCL; defined as limited stage by routine staging criteria in lymphoma involving FDG-PET and bone marrow biopsies (the Lugano criteria)[21]
* Patients with grade 3B follicular lymphoma and transformed indolent lymphoma are included
* Ages ≥ 18
* Measurable disease, assessable by radiographic examination with FDG-PET showing involvement
* Access to archived or fresh/frozen tumor biopsies
* No uncontrolled medical comorbidities
* Adequate cardiac function (EF > or equal to 50%), no unstable angina
* Adequate renal function (GFR > 60)
* Adequate liver function (liver function tests should be no greater than 2 x upper limit of normal) including normal bilirubin levels, no greater than 2 x upper limit of normal unless patient has a history of Gilbert's disease
* Adequate marrow reserves as indicated by complete blood count in the judgment of the treating investigator

Exclusion Criteria:

* Pregnancy, positive serum HCG within 28 days of enrollment, or breast-feeding
* Bulky disease greater than 10 cm in any dimension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between fluorodeoxyglucose positron emission tomography (FDG-PET) and MRD, as measured by circulating tumor plasma DNA (ctDNA) in patients with early stage diffuse large B cell lymphoma (DLBCL). | 5 years

SECONDARY OUTCOMES:
PET CR rate | 5 years
Change in minimal residual disease (MRD) from baseline to time of re-staging PET | 5 years
Re-staging Deauville score of 1, 2, or 3 (negative PET scan) | 5 years
Following 3 cycles of R-CHOP, if PET scan demonstrates complete response, defined by Deauville score of 1, 2, or 3 (negative PET scan), radiation therapy will not be required moving forward | 5 years
Toxicity rates using CTCAE v4.03 | 5 years
Changes in quality of life using PROMIS scale 10 scale will be administered to patients at the time of diagnosis, at the conclusion of all therapy, and at 12 month intervals | 5 years
Overall survival (OS) of patients through two years of follow-up. | Patients will be assessed by physical exam and routine bloodwork every 3 months in the 1st year after conclusion of treatment, and every 6 months in the second year following treatment. They will be assessed yearly during years 3, 4 and 5.
Progression free survival (PFS) | From time of baseline scan through two years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carla Casulo, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided